CLINICAL TRIAL: NCT01801293
Title: A Phase 1 Study to Evaluate the Pharmacokinetics, Metabolism, and Excretion of GS-5806
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-218-0109
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: RSV Infection
Keywords: RSV infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — presatovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Arm (Experimental): One-time single dose of 50 mg radiolabeled GS-5806 administered orally in 3 capsules in the morning.
  Interventions: Drug: GS-5806

INTERVENTIONS:
Drug: GS-5806

SUMMARY:
This is a single center, open-label, Phase 1 study to determine the mass balance of of GS-5806 following administration of a single, oral dose of radiolabeled [14C]-GS-5806 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have a calculated body mass index (BMI) from 19 to 30 kg/m2 at study screening.
* In the opinion of the Investigator, subjects must be in good health based upon medical history, physical examination (including vital signs), and screening and baseline laboratory evaluations (hematology, chemistry, and urinalysis must fall within the normal range of the local laboratory's reference ranges unless the results have been determined by the Investigator to have no clinical significance).
* Agree to utilize a highly effective method of contraception during heterosexual intercourse from baseline throughout the study period and for 90 days following discontinuation of study drug.
* Refrain from sperm donation from Day -1 through completion of the study and continuing for at least 90 days from the date of last dose of study drug.
* Have a creatinine clearance (CLcr) > 80 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at the screening evaluation.
* Anticipated, regular, average bowel movement of 1-2 per day.

Exclusion Criteria:

* Smokers, use of nicotine or nicotine-containing products within 90 days prior to the first dose of study drug. Smokers will be defined as any subject who reports tobacco use and/or who has a urine cotinine ≥200 ng/mL at screening.
* A positive HIV-1 antibody, Hepatitis B surface antigen (HBsAg), or Hepatitis C antibody test result.
* Have any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol.
* Have previously participated in an investigational trial involving administration of any investigational compound within 30 days prior to study dosing.
* Have participated in studies using radiomaterials or ionizing radiations or have been otherwise exposed to significant diagnostic (excluding dental X-rays), therapeutic, or occupational radiation.
* Current alcohol or substance abuse as judged by the Investigator or as determined by a positive alcohol or drug test at screening or baseline visit.
* Have poor venous access and are unable to donate blood.
* Have donated blood within 56 days of study dosing or plasma within 7 days of study dosing.
* Have been vaccinated within 90 days of study dosing or, for the influenza vaccine, within 14 days prior to study dosing.
* Have taken any prescription medications or over-the-counter medications, including herbal products, or medications that affect gastric pH (ie, antacids, H2RAs, and/or proton pump inhibitors) within 28 days of commencing study drug dosing with the exception of vitamins, acetaminophen, and ibuprofen.
* Have taken any systemic steroids, immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents during the study (eg, corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies).
* Evidence of any of the following:

  1. Clinically significant ECG abnormalities.
  2. Syncope, palpitations, or unexplained dizziness.
  3. Liver disease (including known Gilbert's Disease) or clinical evidence of liver injury or hepatic synthetic dysfunction.
  4. Severe peptic ulcer disease, gastroesophageal reflux disease, or other gastric acid hypersecretory conditions requiring prolonged (>6 months) medical treatment.
  5. History of medical or surgical treatment that permanently alters the gastric conditions (eg, gastrectomy).
  6. Significant drug sensitivity or drug allergy.
  7. Known hypersensitivity to sulfa drugs.
  8. Known hypersensitivity to the study drug, metabolites or formulation excipients.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Urine and fecal recovery of total [14C]-radioactivity | 22 days
  The primary outcome measure of this study is the urine and fecal recovery of total [14C]-radioactivity.

SECONDARY OUTCOMES:
Recovery of [14C]-GS-5806 | 22 days
  The secondary endpoint measure is the urine and fecal recovery of [14C]-GS-5806 and, where measurable, its metabolite(s).

OTHER OUTCOMES:
Plasma and blood concentration and PK parameters - Radioactivity | 22 days
  Secondary endpoint measures include the plasma and blood concentration and PK parameters of total [14C]-radioactivity, and the plasma to blood ratio of [14C]-radioactivity.
Plasma and blood concentration and PK parameters - Non-radiolabeled | 22 Days
  Secondary endpoint measures include the plasma concentration and PK parameters of non-radiolabeled GS-5806 and, where measurable, its metabolite(s).
Plasma and blood concentration and PK parameters - [14C]-GS-5806 | 22 Days
  Secondary endpoint measures include the plasma concentration and PK parameters of [14C]-GS-5806, and where measurable, its metabolite(s).

CONTACTS AND LOCATIONS:
Overall Officials: Seth Toback, M.D., Study Director — Gilead Sciences
Locations (1):
- Investigational Site, Madison, Wisconsin, United States